CLINICAL TRIAL: NCT07401082
Title: Postoperative Pain and Quality of Life With Different Modalities of Mesh Fixation in Laparoscopic Trans-Abdominal Pre-Peritoneal Repair of Inguinal Hernia. A Randomized Controlled Trial
Brief Title: Mesh Fixation Methods in Laparoscopic Hernia Repair: Glue vs. Sutures vs. Tacks
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Eid Ali Ahmed Aziz, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS-358-2024
Record Dates: First submitted 2026-01-30; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Inguinal Hernia
Keywords: Inguinal hernia; Laparoscopic Hernia Repair; TAPP; Transabdominal Preperitoneal Repair; Mesh Fixation; Surgical Glue; Cyanoacrylate; Sutures; Tacks; Carolinas Comfort Scale; Postoperative Pain
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative | interventions — tetra-4-amidinophenoxypropane

STUDY DESIGN:
Intervention Model Description: Participants are randomized into one of three parallel groups (glue, sutures, tacks) and remain in that group for the duration of the study. All groups undergo the same surgical procedure (TAPP) with only the mesh fixation method differing.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glue Mesh Fixation (Experimental): Participants in this arm will undergo laparoscopic transabdominal preperitoneal (TAPP) inguinal hernia repair with mesh fixation using a cyanoacrylate-based surgical adhesive (Glubran-2®) applied via a dedicated applicator (GlueTack device). The mesh will be secured with small drops of glue at its corners.
  Interventions: Device: Cyanoacrylate Surgical Adhesive Fixation; Procedure: Laparoscopic Transabdominal Preperitoneal (TAPP) Inguinal Hernia Repair with Polypropylene Mesh Fixation. .
- Suture Mesh Fixation (Experimental): Participants in this arm will undergo laparoscopic transabdominal preperitoneal (TAPP) inguinal hernia repair with mesh fixation using two non-absorbable polypropylene sutures placed at the medial and lateral ends of the mesh. This is a traditional mechanical fixation method.
  Interventions: Procedure: Suture Mesh Fixation; Procedure: Laparoscopic Transabdominal Preperitoneal (TAPP) Inguinal Hernia Repair with Polypropylene Mesh Fixation. .
- Tack Mesh Fixation (Active Comparator): Participants in this arm will undergo laparoscopic transabdominal preperitoneal (TAPP) inguinal hernia repair with mesh fixation using helical titanium tacks (e.g., ProTack®). This is a standard mechanical fixation method commonly used in laparoscopic hernia repair. Tacks are placed around the periphery of the mesh, avoiding critical neurovascular zones.
  Interventions: Device: Helical Titanium Tack Fixation; Procedure: Laparoscopic Transabdominal Preperitoneal (TAPP) Inguinal Hernia Repair with Polypropylene Mesh Fixation. .

INTERVENTIONS:
Device: Cyanoacrylate Surgical Adhesive Fixation — Fixation of the polypropylene mesh using a cyanoacrylate-based surgical adhesive (Glubran-2®). The adhesive is applied in small drops at the mesh corners using a specific applicator device (GlueTack) to secure the mesh to the abdominal wall without mechanical penetration.
  Arms: Glue Mesh Fixation
Procedure: Suture Mesh Fixation — Fixation of the polypropylene mesh using two non-absorbable polypropylene sutures. The sutures are placed laparoscopically at the medial and lateral ends of the mesh to mechanically secure it to the abdominal wall tissues (e.g., Cooper's ligament, transversalis fascia).
  Arms: Suture Mesh Fixation
Device: Helical Titanium Tack Fixation — Fixation of the polypropylene mesh using multiple helical titanium tacks ( ProTack®). The tacks are fired laparoscopically around the periphery of the mesh, penetrating the abdominal wall to mechanically secure the mesh in place, while avoiding anatomical danger zones.
  Arms: Tack Mesh Fixation
Procedure: Laparoscopic Transabdominal Preperitoneal (TAPP) Inguinal Hernia Repair with Polypropylene Mesh Fixation. . — All participants in this study will undergo Laparoscopic Transabdominal Preperitoneal (TAPP) Repair of Inguinal Hernia, which is the standard surgical procedure. This minimally invasive technique involves:
  Creation of Pneumoperitoneum: The abdominal cavity is inflated with carbon dioxide gas.
  Port Placement: Three small incisions are made for camera and instrument ports.
  Peritoneal Incision: The peritoneum (inner abdominal lining) is cut to access the preperitoneal space in the groin.
  Hernia Reduction: The hernia sac and contents are pushed back into the abdominal cavity.
  Mesh Placement: A synthetic polypropylene mesh is positioned to cover the entire myopectineal orifice (the weak area where hernias occur).
  Mesh Fixation: The mesh is secured using one of three study methods (glue, sutures, or tacks) according to the assigned intervention arm.
  Peritoneal Closure: The initial peritoneal incision is closed over the mesh to isolate it from the abdominal organs.

SUMMARY:
This study is a clinical trial that aims to compare three different methods for securing a surgical mesh during a specific type of groin (inguinal) hernia repair surgery. The surgery is performed using a minimally invasive, keyhole technique called TAPP.

The main questions this study aims to answer are:

Which mesh fixation method-surgical glue, stitches (sutures), or small metal coils (tacks)-results in less pain for patients after surgery?

Which method leads to a better quality of life and less feeling of the mesh inside the body after recovery?

Is there a difference in how long the surgery takes with each method?

To answer these questions, researchers will compare the three methods to see which one works best for patient comfort and recovery.

Adults aged 21-60 years with a new inguinal hernia who are having laparoscopic TAPP surgery can participate.

Participants will be randomly assigned to one of three groups:

Group 1: Their mesh will be secured using surgical glue.

Group 2: Their mesh will be secured using stitches (sutures).

Group 3: Their mesh will be secured using small metal coils (tacks).

All other parts of the surgery and care after surgery will be the same.

Participants will:

Have the laparoscopic TAPP hernia repair surgery.

Report their pain levels after surgery using a simple scale.

Answer questions about their comfort and quality of life during follow-up visits at 1, 3, and 6 months after surgery.

DETAILED DESCRIPTION:
This study is a prospective, single-center, randomized controlled trial designed to compare the postoperative outcomes associated with three distinct mesh fixation modalities in laparoscopic Trans-Abdominal Pre-Peritoneal (TAPP) inguinal hernia repair.

Scientific Rationale:

While mesh reinforcement has drastically reduced recurrence rates in hernia surgery, chronic postoperative pain and mesh-related discomfort remain significant concerns that impact patient quality of life. The method of securing the mesh is hypothesized to be a key factor influencing these outcomes. Mechanical fixation with tacks or sutures may cause tissue trauma or nerve irritation, whereas adhesive fixation provides an atraumatic alternative. Direct comparative data on these three common techniques(glue, sutures, and tacks) within the standardized TAPP procedure is limited.

Study Design:

A total of 75 eligible participants will be enrolled and equally randomized into one of three parallel intervention arms in a 1:1:1 ratio. The randomization sequence will be computer-generated. Due to the nature of the interventions, blinding of the surgeon is not feasible; however, outcome assessors and the statistician will be blinded to group assignment where possible.

Interventional Protocol:

All participants will undergo a standardized TAPP procedure under general anesthesia. After creation of the preperitoneal space and placement of a polypropylene mesh over the myopectineal orifice, fixation will be performed according to the assigned group:

Glue Fixation Group: Fixation using a cyanoacrylate-based surgical adhesive (e.g., Glubran-2®) applied with a specific applicator.

Suture Fixation Group: Fixation using two non-absorbable polypropylene sutures placed at the medial and lateral ends of the mesh.

Tack Fixation Group: Fixation using helical titanium tacks (e.g., ProTack®), with careful avoidance of the "triangle of doom" and "triangle of pain" anatomical zones.

Follow-up and Assessments:

Participants will be followed for a period of six months postoperatively. Structured assessments will occur at designated intervals:

Pain Assessment: Measured using the Visual Analogue Scale (VAS) on postoperative day 1 and at 1, 3, and 6 months.

Quality of Life and Mesh Sensation: Assessed using the Carolinas Comfort Scale (CCS), a validated hernia-specific questionnaire, at 1, 3, and 6 months.

Clinical Outcomes: Operative time, length of hospital stay, time to return to normal work/activities, incidence of complications (seroma, hematoma, infection), and hernia recurrence will be systematically recorded.

Statistical Analysis:

Data will be analyzed on an intention-to-treat basis. Continuous variables will be compared using ANOVA or Kruskal-Wallis tests as appropriate, followed by post-hoc pairwise comparisons. Categorical variables will be analyzed using the Chi-square or Fisher's exact test. A p-value of <0.05 will be considered statistically significant.

Study Significance:

This trial aims to provide high-level evidence to guide surgical practice by identifying the mesh fixation technique associated with the most favorable balance of reduced postoperative pain, improved quality of life, and cost-effectiveness, without compromising the durability of the repair.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21 to 60 years
* Diagnosis of primary (de novo) inguinal hernia
* Hernia type: unilateral or bilateral, direct or indirect
* Scheduled for elective laparoscopic transabdominal preperitoneal (TAPP) repair
* Able to provide informed consent

Exclusion Criteria:

* Age <21 or >60 years
* Recurrent inguinal hernia
* Complicated hernia (irreducible, incarcerated, obstructed, or strangulated)
* Contraindication to laparoscopic surgery or general anesthesia
* Significant comorbid conditions making surgery high-risk (ASA class ≥III)
* Chronic pain syndrome or regular use of strong analgesics
* Allergy to mesh materials (polypropylene) or fixation components (cyanoacrylate, titanium)
* Participation in another clinical trial
* Inability to complete follow-up or comply with study protocol

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | Assessed on postoperative Day 1 and at 1 month, 3 months, and 6 months postoperatively.
  Intensity of pain measured using the Visual Analogue Scale (VAS), a 10-point scale where 0 = no pain and 10 = worst pain imaginable.
Postoperative Quality of Life and Mesh Sensation | Assessed at 1 month, 3 months, and 6 months postoperatively.
  Patient-reported quality of life and mesh-related symptoms were measured using the Carolinas Comfort Scale (CCS), a validated hernia-specific outcome measure. The CCS consists of 23 items evaluating pain, mesh sensation, and movement limitation during daily activities, each scored from 0 (no symptoms) to 5 (disabling symptoms), yielding a total score range of 0-115. Higher scores indicate worse postoperative comfort and quality of life.
Operative Time | Recorded on the day of surgery.
  Total duration of surgery, measured from skin incision to skin closure (in minutes).

SECONDARY OUTCOMES:
Hernia Recurrence | Assessed at 6 months postoperatively.
  Clinical or radiological evidence of recurrent inguinal hernia at the operated site.
Time to Return to Work/Normal Activity | Assessed within the first 4 weeks postoperatively.
  Number of days from surgery until the patient returns to their regular employment or daily activities.
Length of Hospital Stay | Measured during the immediate postoperative period (typically 1-2 days).
  Number of days from surgery to discharge from the hospital.
Postoperative Complications | Assessed on postoperative Day 1 and at 1 month, 3 months, and 6 months postoperatively
  Incidence of surgical complications including seroma, hematoma, wound infection, mesh infection, and scrotal edema.
Direct Material Cost of Mesh Fixation Device | Recorded on the day of surgery.
  The direct material cost of the specific fixation device used in each study arm is recorded in US Dollars (USD). Costs are categorized into three predetermined ranges based on hospital procurement prices: Low ($30-60), Moderate ($200-300), and High ($350-500). Data will be aggregated and reported as the proportion of participants in each study arm falling into these cost categories.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Eid Aziz, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Al-Manial Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No